CLINICAL TRIAL: NCT06868797
Title: Acute Reno-Cardiac Action of Dapagliflozin In Advanced Heart Failure Patients on Heart Transplant Waiting List
Acronym: ARCADIA-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BAUDRY Guillaume, coordinating investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023PI024; 2024-A02450-47 (Other: ID-RCB)
Record Dates: First submitted 2025-02-17; First posted 2025-03-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients followed for end-stage heart failure (Other): Patients followed for end-stage heart failure and waiting for heart transplantation. This cohort will focus on cardio-renal assessment of advanced HF patients treated with optimal pharmacologic therapy including dapagliflozin. The biological material and clinical data collected will allow us to better understand the advanced HF and to generate new research hypotheses.
  Interventions: Other: Biological sample for the measurement of suPAR levels.

INTERVENTIONS:
Other: Biological sample for the measurement of suPAR levels. — Biological sample for the measurement of plasminogen activator receptor (suPAR) level at baseline and at 6 months follow up to assess the evolution of cardio-renal interaction in HF patients listed for heart transplant treated by GDMT including dapagliflozin.

SUMMARY:
Heart failure affects 1 to 2% of the adult population in developed countries, representing about 55 million people worldwide.

Advanced heart failure is a condition where the heart can no longer provide sufficient cardiac output or equilibrate pressures within its chambers, leading to symptoms such as shortness of breath, fatigue, and water and salt retention.

Heart failure affects the kidneys by reducing blood flow directed to them, sometimes leading to kidney congestion. In the long term, this can degrade kidney function. Common medications used to treat heart failure, such as diuretics, can sometimes worsen kidney failure. This link between the heart and the kidneys is known as cardio-renal syndrome and requires careful management of both organs to prevent mutual degradation.

Dapagliflozin is an SGLT2 inhibitor medication used to treat type 2 diabetes, heart failure, and certain kidney diseases. It helps reduce blood sugar, improve heart and kidney function, while promoting the elimination of excess salt and water.

However, there are limited data regarding the progression of cardio-renal interactions in patients with advanced heart failure. Yet, advanced heart failure is often associated with kidney dysfunction.

The protein called suPAR is found in the blood of patients developing kidney disease and/or during the onset of acute kidney injury. This protein will allow to characterize a population of patients with advanced heart failure receiving optimized medical treatment, including dapagliflozin.

The main objective of this research is to assess, based on the suPAR protein level in the blood, the progression of cardio-renal damage between inclusion and 6 months in patients with advanced heart failure who are listed for a heart transplant and treated with a therapy including dapagliflozin.

The study plans 5 visits over 12 months. The research will take place in the cardiology department of several French hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 85 years
2. NYHA class ≥3
3. LVEF ≤ 35%
4. On GDMT (including dapagliflozin) based on current heart failure practice guidelines at maximal tolerated dose
5. On waiting list (or on the registration pathway) for heart transplantation after multidisciplinary Heart Team decision, with anticipated access to heart transplant ≥ 6 months or in a pre-transplant pathway.
6. Person affiliated to a social security scheme or beneficiary of such a scheme.
7. A person who has received full information about the organization of the clinical research and has signed an informed consent form.

Exclusion Criteria:

1. Priority patient on waiting list for heart transplantation.
2. Etiology of heart failure due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy.
3. Inotrope dependent, existence of ongoing mechanical circulatory support
4. Current acute decompensated HF or hospitalization due to decompensated HF <30 days prior to the enrolment.
5. History of any organ transplant or prior implantation of a ventricular assistance device (VAD) or similar device, or implantation expected after inclusion.
6. Any recent interventional procedure likely to improve symptoms and heart failure status (coronary revascularization, percutaneous mitral valve intervention, cardiac resynchronization therapy) < 60 days.
7. Glomerular filtration rate <25 ml/min/1.73 m2, according to CKD-EPI formula
8. Unstable or rapidly progressing renal disease (autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or ANCA-associated vasculitis).
9. Type 1 diabetes mellitus.
10. Participation in another clinical interventional trial.
11. Any condition other than heart failure that could limit survival to less than 12 months.
12. Pregnant women or breastfeeding mothers
13. vulnerable persons (guardianship, curatorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-12 (Estimated)

PRIMARY OUTCOMES:
the change in soluble urokinase-type plasminogen activator receptor (suPAR) levels (ng/ml) | baseline and 6 months of follow-up.
  the change in soluble urokinase-type plasminogen activator receptor (suPAR) levels (ng/ml) between the baseline and 6 months of follow-up.

SECONDARY OUTCOMES:
VO2 max | baseline and 6 months of follow-up.
  Functional status at baseline and 6 months assessed by VO2 max assessment
Delta GFR estimated by CKD-EPI formula (ml/min/1.73m²) | baseline and 6 months of follow-up.
  The following parameters are collected at baseline to identify predictive factors associated with secondary endpoint. These parameters should not be considered as endpoints themselves:
  * Hemodynamic Parameters: cardiac output (L/min), pulmonary capillary wedge pressure (mmHg), pulmonary artery systolic and mean pressure (mmHg), right atrial pressure (mmHg).
  * Echocardiographic Parameters: LVEF (%), mitral regurgitation grade (0-4), left atrial volume (mL /m2).
  * Biological Parameters: Nt-proBNP (ng/L), Creatinine (µmol/L), GFR evaluate by Iohexol clearance (ml/min) or other method (ml/min) (inuline, EDTA chrome51 (51Cr EDTA), Iothalamate clearance),plasma volume calculated from haemoglobin (g/L) and haematocrit,(%) bilirubin (µmol/L), AST (UI/L), ALT (UI/L), kalemia (mmol/L), cystatin C (mg/L), sST2 (ng/mL), gremlins 1(pg/mL), FGF 23 (C terminal and intact) (pg/mL).
  * Congestion Markers: Clinical, biological, echocardiographic, and hemodynamic markers.
Rate of composite outcome (hospitalization for acute heart failure or all cause death). | 6 months of follow-up.
  The following parameters are collected at baseline to identify predictive factors associated with secondary endpoint. These parameters should not be considered as endpoints themselves:
  * Hemodynamic Parameters: cardiac output (L/min), pulmonary capillary wedge pressure (mmHg), pulmonary artery systolic and mean pressure (mmHg), right atrial pressure (mmHg).
  * Echocardiographic Parameters: LVEF (%), mitral regurgitation grade (0-4), left atrial volume (mL /m2).
  * Biological Parameters: Nt-proBNP (ng/L), Creatinine (µmol/L), GFR evaluate by Iohexol clearance (ml/min) or other method (ml/min) (inuline, EDTA chrome51 (51Cr EDTA), Iothalamate clearance),plasma volume calculated from haemoglobin (g/L) and haematocrit,(%) bilirubin (µmol/L), AST (UI/L), ALT (UI/L), kalemia (mmol/L), cystatin C (mg/L), sST2 (ng/mL), gremlins 1(pg/mL), FGF 23 (C terminal and intact) (pg/mL).
  * Congestion Markers: Clinical, biological, echocardiographic, and hemodynamic markers.
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | baseline and 12 months.
  Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ total symptom score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Global Leadership Initiative on Malnutrition criteria (GLIM Criteria) | baseline and 6 months
  To assess changes in nutritional status according to Global Leadership Initiative on Malnutrition criteria status between Baseline and 6 months. Categories : no malnutrition, moderate malnutrition, or severe malnutrition
Daily food and nutrient intake | baseline or the month following baseline
  The food frequency questionnaire evaluate the frequency of consumption and portion size for 170 foods, we then calculate the daily food intake (in g/day). Nutritrional values are determined by converting food intake into nutrient intake using a french food composition table. Each item can have a minimum intake of 0, with quantities varying based on the specific food and individual consumption.
cardiovascular death | 12 months
  To assess incidence of cardiac and renal adverse events.
unplanned hospitalization for Heart failure | 12 months
  To assess incidence of cardiac and renal adverse events. The definition for unplanned heart failure hospitalization requires: 1) a hospital stay for worsening heart failure for >24 h; and 2) administration of intravenous or mechanical heart failure therapies, especially loop diuretics 3) heart failure symptoms/signs.
worsening of Heart failure | 12 months
  To assess incidence of cardiac and renal adverse events. The definition for worsening of heart failure requires an administration of loop diuretics intravenous (ambulatory or home-care) due to a worsening of heart failure symptoms/signs.
cardiac transplantation | 12 months
  To assess incidence of cardiac and renal adverse events
ECMO | 12 months
  To assess incidence of cardiac and renal adverse events
Left Ventricular Assist Device | 12 months
  To assess incidence of cardiac and renal adverse events
Delisting from national waiting list | 12 months
  to assess incidence of cardiac and renal adverse events
renal death | 12 months
  To assess incidence of cardiac and renal adverse events.
chronic dialysis | 12 months
  To assess incidence of cardiac and renal adverse events.
renal transplantation | 12 months
  To assess incidence of cardiac and renal adverse events.
End stage renal disease | 12 months
  To assess incidence of cardiac and renal adverse events. Chronic dialysis, renal transplantation or sustained eGFR <15 mL/min/1.73m²
worsening cardio-renal syndrome | 12 months
  To assess incidence of cardiac and renal adverse events. Worsening cardio-renal syndrome was defined according to the Kidney Disease Improving Global Outcomes (KIDGO) criteria as a ≥ 26.5 µmol/L (0.3mg/dL) increase in serum creatinine or 1.5-1.9 times baseline increase in serum creatinine or a urine output <0.5 ml/kg/h for 6-12 hours.
GFR estimated by CKD-EPI formula (serum creatinine cystatin or both) | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR.
GFR estimated by MDRD formula | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR.
urinary creatinine (renal functional assessment (BFR)) | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR.
iohexol clearance | baseline and 6 months
  to assess the degree of agreement between the different methods of estimating GFR
inuline clearance | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR
EDTA chrome51 | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR
Iothalamate clearance | baseline and 6 months
  To assess the degree of agreement between the different methods of estimating GFR
PLAUR gene expression | baseline and 6 months
  To assess the change in gene expression (including PLAUR gene) using the RNA collected at baseline and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GIRERD, MD-PhD, Study Chair — CHRU de NANCY
Locations (11):
- France (11):
  - Hospice Civil de Lyon - Hôpital Louis PRADEL, Bron
  - CHU Grenoble, La Tronche
  - CHU Montpellier, Montpellier
  - Chu Nantes, Nantes
  - Aphp Hegp, Paris
  - CHU Bordeaux, Pessac
  - CHU Rennes, Rennes
  - Chu Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Chru Nancy, Vandœuvre-lès-Nancy